CLINICAL TRIAL: NCT05647343
Title: A Phase I, Double-blind, Randomized, Placebo-controlled Study to Assess the Safety and Pharmacokinetics of ATL-001 (Ciclopirox Olamine) in Healthy Volunteers
Brief Title: Study to Assess the Safety and Pharmacokinetics of ATL-001 (Ciclopirox Olamine) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Atlas Molecular Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: ATL001-PI-CEP
Record Dates: First submitted 2022-11-22; First posted 2022-12-12 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Adverse Effect of Drugs and Medicaments in Therapeutic Use
MeSH Terms: interventions — Ciclopirox

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- ATL-001 0.2 mg/kg vs Placebo (Experimental): Cohort 1: ATL-001 at 0.2 mg/kg or Placebo (depending on randomization) will be administered during 5 days
  Interventions: Drug: Ciclopirox Olamine Oral; Other: Placebo
- ATL-001 0.5 mg/kg vs Placebo (Experimental): Cohort 2: ATL-001 at 0.5 mg/kg or Placebo (depending on randomization) will be administered during 5 days
  Interventions: Drug: Ciclopirox Olamine Oral; Other: Placebo
- ATL-001 1 mg/kg vs Placebo (Experimental): Cohort 3: ATL-001 at 1 mg/kg or Placebo (depending on randomization) will be administered during 5 days
  Interventions: Drug: Ciclopirox Olamine Oral; Other: Placebo
- ATL-001 2 mg/kg vs Placebo (Experimental): Cohort 4: ATL-001 at 2 mg/kg or Placebo (depending on randomization) will be administered during 5 days
  Interventions: Drug: Ciclopirox Olamine Oral; Other: Placebo
- ATL-001 4 mg/kg vs Placebo (Experimental): Cohort 5: ATL-001 at 4 mg/kg or Placebo (depending on randomization) will be administered during 5 days
  Interventions: Drug: Ciclopirox Olamine Oral; Other: Placebo

INTERVENTIONS:
Drug: Ciclopirox Olamine Oral — On the morning of Day 1 to Day 5, each participant will receive a single oral dose of ATL-001 or placebo
Other: Placebo — On the morning of Day 1 to Day 5, each participant will receive a single oral dose of ATL-001 or placebo

SUMMARY:
The goal of this clinical trial is to assess the safety, tolerability and pharmacokinetics of ATL-001 (ciclopirox olamine) in healthy volunteers

DETAILED DESCRIPTION:
Participants will receive either the investigational drug (ATL-001) or Placebo (inactive substance). Neither the participant nor the Investigator will know to which of these study drug groups each participant has been assigned. In case of an emergency, however, the Investigator can get this information.

After a 30-day Screening period to confirm the eligibility, the prticipants will be treated for 5 days (the treatment period) and followed by 30 days of observation and assessment of treatment outcomes (the follow-up period).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subjects 18 to 65 years of age, inclusive
2. Body mass index (BMI) within the range of 18.0 to 33.0 kg/m2, inclusive, and a minimum weight of at least 50.0 and maximum weight of 100.0 kg at Screening
3. Estimated Glomerular Filtration Rate (eGFR) > 90 mL/min/1.73 m2 at Screening
4. Female subjects of childbearing potential must be using and willing to continue using two medically acceptable contraceptive precautions from Screening and for at least 1 month after the last study drug administration. Medically acceptable forms of contraception include sexual abstinence [periodic abstinence (e.g., calendar, ovulation, symptothermal and post-ovulation methods) are not acceptable], combined (oestrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal or transdermal), intrauterine devices (IUD), intrauterine hormone-releasing systems, and bilateral tubal ligation for subjects
5. Female subjects of non-childbearing potential must be amenorrhoeic for at least 2 years or had a hysterectomy and/or bilateral oophorectomy/salpingo-oophorectomy (as determined by subject medical history)
6. Male subjects of reproductive potential with a partner(s) of childbearing potential must be using and willing to continue using two medically acceptable contraceptive precautions from Screening and for at least 1 month after the last study drug administration. Medically acceptable forms of contraception include abstinence, vasectomy, or male condom for subjects
7. Female subjects must have a negative pregnancy test
8. Must understand and provide written informed consent prior to the initiation of any protocol-specific procedures
9. Must be willing and able to abide by all study requirements and restrictions

Exclusion Criteria:

1. Current drug or alcohol dependence (excluding caffeine), based on self-report, including subjects who have been in a drug rehabilitation program
2. Current smoker or a history of using tobacco products within 3 months prior to Screening
3. Clinically significant abnormalities on physical examination, medical history, 12-lead ECG (i.e., QTc > 440 ms for male subjects and > 450 ms for female subjects), vital signs, or laboratory values, as judged by the investigator or designee
4. History or presence of any clinically significant illness (e.g., cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, oncologic, musculoskeletal, or psychiatric) or any other condition, which in the opinion of the investigator would jeopardize the safety of the subject or the validity of the study results
5. Use of a non-prescription drug within 14 days prior to the first drug administration. Subjects who have taken over-the-counter medication may still be entered into the study, if in the opinion of the investigator or designee, the medication received will not interfere with the study procedures or data integrity or compromise the safety of the subject
6. Use of any prescription medications, recreational drugs, or natural health products (except vitamin or mineral supplements, acceptable forms of birth control, and hormone replacement) within 14 days prior to first drug administration or throughout the study, unless in the opinion of the investigator or designee, the product will not interfere with the study procedures or data integrity or compromise the safety of the subject
7. Use of any medication that interfere with the glucuronidation metabolic pathway within 14 days prior to first drug administration
8. Positive urine drug screen
9. Positive breath alcohol test. If a subject presents with positive breath alcohol test, the subject may be rescheduled at the discretion of the investigator or designee
10. Female subjects who are currently pregnant or lactating or who are planning to become pregnant within 60 days of last study drug administration
11. Known history of allergy or hypersensitivity to any component of the active drug or placebo
12. Positive for Hepatitis B, Hepatitis C, HIV or COVID-19
13. Treatment with any investigational drug within 30 days prior to first drug administration in the treatment phase
14. A subject who, in the opinion of the investigator or designee, is not considered to be suitable and is unlikely to comply with the study protocol for any reason

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-03-31 (Actual); Primary Completion 2024-04-08 (Actual); Study Completion 2024-04-08 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | 3.5 months, with up to 66 days per participant
  Incidence of adverse events (AEs) and of clinically relevant changes in vital signs values, electrocardiogram (ECG) data, physical examination and laboratory safety data for four different doses of ATL-001

SECONDARY OUTCOMES:
Derived pharmacokinetic parameters for ATL-001 | 6 days per participant
  Area under the plasma drug concentration
Derived pharmacokinetic parameters for ATL-001 | 6 days per participant
  Time curve (AUC(0-last), AUC(0-12), AUC(0-24))
Derived pharmacokinetic parameters for ATL-001 | 6 days per participant
  Maximum observed plasma drug concentration (Cmax)
Derived pharmacokinetic parameters for ATL-001 | 6 days per participant
  Time to maximum observed plasma drug concentration (tmax)
Derived pharmacokinetic parameters for ATL-001 | 6 days per participant
  Apparent terminal half-life (t1/2)
Derived pharmacokinetic parameters for ATL-001 | 6 days per participant
  Apparent total body clearance (CL/F)
Derived pharmacokinetic parameters for ATL-001 | 6 days per participant
  Apparent volume of distribution (Vz/F)

CONTACTS AND LOCATIONS:
Locations (1):
- Hassman Research Institute, LLC, Berlin, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2023-12-13): https://cdn.clinicaltrials.gov/large-docs/43/NCT05647343/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-26): https://cdn.clinicaltrials.gov/large-docs/43/NCT05647343/SAP_001.pdf